CLINICAL TRIAL: NCT04126421
Title: Vitamin E Stabilized Highly Cross-linked Polyethylene in Reversed Hybrid Total Hip
Brief Title: Vitamin E Polyethylene in Semented Cups
Acronym: E1vsMar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Peder Svenkerud Thoen, MD, Consultant Orthopedic Surgery, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010/2621a
Record Dates: First submitted 2019-09-29; First posted 2019-10-15 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Total Hip Arthroplasty (THA)
Keywords: Highly cross-linked polyethylene (HXLPE); Vitamin E infused polyethylene

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT). Randomized to either E1 semented cup or Marathon semented cup in total hip arthroplasty (THA).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E1 Vitamin E infused HXLPE (Active Comparator): E1 Vitamin E infused highly cross-linked polyethylene (HXLPE)
  Interventions: Device: Prosthesis component (acetabular cup) E1 cup
- Marathon HXLPE (Active Comparator): Marathon highly cross-linked polyethylene (HXLPE)
  Interventions: Device: Prosthesis component (acetabular cup) Marathon cup

INTERVENTIONS:
Device: Prosthesis component (acetabular cup) E1 cup — Semented acetabuar cup With E1 cup
  Other Names: E1 cup
  Arms: E1 Vitamin E infused HXLPE
Device: Prosthesis component (acetabular cup) Marathon cup — Semented acetabuar cup With Marathon cup
  Other Names: Marathon cup
  Arms: Marathon HXLPE

SUMMARY:
A prospective randomized controlled study evaluating the wear and migration of cemented acetabular sockets with third generation highly cross-linked vitamin E infused polyethylene and second generation highly crosslinked UHMWPE using Radiostereometric Analysis (RSA).

DETAILED DESCRIPTION:
Background Reducing the rate of polyethylene (PE) wear in acetabular sockets and thereby increasing the lifespan of Total Hip Arthroplasty (THA) has been a major concern in the orthopaedic community for decades. Wear of PE and osteolysis followed by late aseptic loosening of the prosthesis is the main reason for revision surgery after THA in Norway.

During 2008 in Norway 805 out of a total of 1114 revised THA were subjugated to surgery due to aseptic loosening or osteolysis without loosening. The DRG (Diagnose Related Grouping) weight is 5.49 for secondary THA and every DRG point has a value of 33.647 NOK adding up to a direct total cost for revision after aseptic loosening of approximately 27 million USD.

Caput prosthesis with a diameter of 32mm or more has the major advantage to increase the Range of Motion (ROM) and to reduce the risk of dislocation of the hip but, the larger the caput prosthesis the more adhesive wear can be expected. This and the relative failure of metal on PE gave the incentive to develop and take into clinical practise bearings with increased resilience to wear. Today, there exists a wide range of options with a substantially lower rate of volumetric wear compared to conventional PE. The biological and immunological in vivo response to wear particles is very complicated and only partially understood. It is clear that host response to wear particles and the corrosion products play a major role in osteolysis around the prosthesis. For metal-on-metal (MoM) bearings the volumetric wear is a magnitude less but the number of particle debris is massively increased. MoM also have the problem with possible teratogen effect and allergy or hypersensitivity side effects. Ceramic on ceramic (cer-cer) has the lowest wear rate of any artificial articulations, but it is still possible to detect biologically active debris particles. Cer-cer also has other challenges including fracture of prosthesis, squeaking hip, narrow margins for placing components and cost.

Polyethylene is a thermoplastic polymer consisting of long chains of the monomer ethylene (C2H4). The mechanical properties of PE depend on variables such as the extent and type of branching and the crystal structure etc.

To improve the wear resistance of the PE an increase in the cross-linking between the chains of polyethylene can be achieved by exposing it to high-energy irradiation. The irradiation also increases the unpaired free electrons (free radicals). Free radicals can react with oxygen and start a chain reaction causing an oxidative degradation of the polyethylene and consequently cause increased wear. 1st generation HXLPE sockets have reduced the mid term incidence of particle-induced osteolysis but retrieved failed first-generation HXLPE sockets have shown surface cracking and signs of in vivo oxidative degradation.

In order to enhance the resistance to mechanical fatigue and reduce oxidative potential 2nd generation HXLPE was developed. To reduce the oxidative potential the polyethylene can be remelted or annealed. Remelting aggravates the mechanical properties of the polyethylene and after annealing there are still remaining free radicals capable of oxidation in vivo. By binding to unpaired free electrons Vitamin E is a scavenger of free radicals. Vitamin E is hydrophobic and can thereby be infused into polyethylene. 3rd generation HXLPE is manufactured below the melting temperature to maintain its mechanical properties and contains Vitamin E to stabilize free radicals. Uncemented Acetabular HXLPE sockets have been shown to have substantially reduced volumetric wear and excellent clinical mid-term results with this type of PE. In Scandinavia the majority of sockets are cemented. The different principles of biological or mechanical stability affects the properties of the socket typically different E-module and the surrounding interface between implant and bone. Conventional PE cemented cups have performed better with less aseptic loosening than uncemented cups. However, as the mechanical properties are changed in highly cross-linked Polyethylene cups, it is not clear whether the higher elasticity of the bone-cement-polyethylene compound might lead to fractures of the more brittle polyethylene. It is therefore not possible to extrapolate clinical results and wear rates from uncemented cups to cemented ones.

Placement of the cup is a crucial parameter for wear and cup survival. Malchau et al. has shown that even high volume surgeons achieve suboptimal placement in 40% of cases. This may depend on patient positioning perioperative, surgical instruments or technique. It is not known whether the surgeon's subjective operative technique directly corresponds to the postoperative evaluation of the cups position. However, adequate cup positioning is crucial in the evaluation of wear. CT is the best method to judge cup position postoperatively and detect osteolysis in the long time perspective.

To the investigators knowledge no randomized controlled study of cemented 3rd generation HXLPE cups utilizing RSA has been conducted.

Hypothesis There is a mid term in vivo reduction of volumetric polyethylene wear with cemented acetabular socket 3rd generation E1™ HXLPE compared with 2nd generation HXLPE.

Material: 70 eligible patients will be included following written informed consent. The participants will be randomized by the envelope method to either E1™ or Marathon™ cemented acetabular socket. The surgery will be performed at the hospitals in Vestre Viken HF and Oslo University hospital HF, Ullevål ortopeden.

Implant The investigators will use two different cemented all PE acetabular sockets;

1. MarathonTM is a 1st generation HXLPE. The polyethylene is cross-linked with 5 Mrad that corresponds to a semi cross-linked PE.
2. The E1™ cemented is an all PE Vitamin E stabilized 3rd generation highly crosslinked UHMWPE. In vitro tests have shown a 99 % decreased volumetric wear rate comparing E1™ with ArComXL™ HXLPE, (highly crosslinked polyethylene) under high contact stress and a 95% reduction in wear rate comparing E1™ with ArCom™ under high contact area stress. Wear particle morphology of E1™ is similar to that of the ArCom™ material.

Collared Corail™ (De Puy, Warsaw, Indiana, USA) uncemented femoral prosthesis is a titanium tapered implant fully coated with 150 micron hydroxyapatite with over 95% survival after 15 years. The caput prosthesis used is the Cobalt Chrome 32 mm Articul/EZE™ (De Puy, Warsaw, Indiana, USA) Refobacin ™ (Biomet Europe, Berlin, Germany) Bone Cement R is a high viscosity, x-ray positive bone cement. A sachet of 40 g Refobacin® Bone Cement R contains 0.5 g gentamicin.

Surgical technique The patient is operated in the position after surgeon's preference and under spinal anaesthesia. Accordingly the approach is after surgeon's preference. When posterolateral approach is chosen a repair of the capsule and the external rotators should be performed. Peroperatively a total of 6 1,0mm tantalum beads are implanted in the perimeter of the socket and 7 beads in the acetabulum. The acetabular socket is positioned as close to 45◦ abduction and 30◦ anteversion as possible.

The surgeon will postoperative directly grade cup position subjectively as anteverted, neutral, retroverted, proximalized, distalized.

Postoperative training Postoperatively the patient is mobilized with full weight bearing from day one.

Radiological analyses Conventional x-ray of pelvis, anterioposterior and lateral projections of hip preoperatively, postoperatively and at 24 (60, 120) months RSA (Radiostereometric analysis) postoperatively, 3, 12, 24 (60, 120) months, the RSA will be analysed at Ullevål University Hospital

Clinical Control Harris Hip Score, EQ-5D and WOMAC will be filled out preoperatively and at 2, 5 and 10 years.

Analysis of data RSA analysis will be performed at the Centre of Implant and Radiostereometric Research Oslo (CIRRO).

The study analysis is conducted under the guidance of CIRRO.

Storage of data Data will be collected and stored at the server for research at Oslo University Hospital. All data is stored anonymously. Each patient receives a study ID. The randomisation key and identity is stored separately.

Statistics Penetration of more than 0,1 mm annually in polyethylene articulations indicates a wear rate that will lead to future osteolysis1.

Scientific value Firstly, if recently developed manufacturing techniques of polyethylene can be shown to decrease the wear rate in vivo, and otherwise have a good clinical and radiological outcome, we have the reason to believe we have the possibility of significantly reducing the revision rate after THA.

Secondly, new implants should thoroughly be investigated and documented before widespread use. This could save many patients from possible disastrous failures as the past has taught us (Boneloc, Carbon compressed Poly).

Safety for the patient. The investigators will follow the normal routines for THA pre, per and postoperatively. Standardized routines in regards to infection and thrombosis prophylaxis following the recommendations from the Norwegian national board of orthopaedics will be followed. Implantation of Tantalum beads has been shown to have negligible side effects.

The E1TM and Marathon PE is clinically tested in uncemented THA, the other components of the prosthesis has more than 10 years clinical and RSA documentation.

Biomet will cover expenses including:

Extra cost of purchasing and storing prosthesis compared with standard prosthesis. Biomet or Stryker has no copy right or any other form of ownership to the result of this study.

ELIGIBILITY:
Inclusion Criteria:

* patients under the age of 75 with primary or secondary arthrosis scheduled for total hip arthroplasty.

Exclusion Criteria:

* a major anatomical deviation, immunosuppressive medication or a significant systemic disease.

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Migration of prothesis components | 5 years
  Migration of prothesis components using radiosterometric analysis of hip x-rays (RSA)

SECONDARY OUTCOMES:
HHS (Patient reported outcome measure (PROMs)) | 10 years
  Harris Hip Score (scale from 0-100, 100 being the best score/result)
EQ-5D (Patient reported outcome measure (PROMs)) | 10 years
  EQ-5D (5 health status descriptions (mobility, self-care, usual activites, pain/discomfort, anxiety/depression) rated by 3 level scale for all categories (1=no problems, 2=moderate problems, 3=extreme problems), in addition there is a health evaluation by VAS scale 0-100, 100 being the worst)
WOMAC (Patient reported outcome measure (PROMs)) | 10 years
  WOMAC (5 items for pain 0-20 (higher score being worse), 2 for stiffness 0-80 (higher score being worse), 17 for functional outcomes 0-68 (higher score being worse))
VAS pain (Patient reported outcome measure (PROMs)) | 10 years
  Visual analog scale (VAS) for pain (scale from 0-10, 10 being the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M Röhrl, PhD, MD, Study Chair — Division of Orthopedic Surgery, Oslo University Hospital
Locations (1):
- Division of Orthopedic Surgery, Oslo Univsersity Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Digas G, Karrholm J, Thanner J, Malchau H, Herberts P. The Otto Aufranc Award. Highly cross-linked polyethylene in total hip arthroplasty: randomized evaluation of penetration rate in cemented and uncemented sockets using radiostereometric analysis. Clin Orthop Relat Res. 2004 Dec;(429):6-16. PMID 15577460
- [Background] Kjærsgaard-Andersen 2010 Orthopaedics today
- [Background] The Norwegian Arthroplasty Register, 2009
- [Background] Garcia-Cimbrelo E, Munuera L. Early and late loosening of the acetabular cup after low-friction arthroplasty. J Bone Joint Surg Am. 1992 Sep;74(8):1119-29. PMID 1400540
- [Background] Barrack RL, Folgueras A, Munn B, Tvetden D, Sharkey P. Pelvic lysis and polyethylene wear at 5-8 years in an uncemented total hip. Clin Orthop Relat Res. 1997 Feb;(335):211-7. PMID 9020220
- [Background] Tarasevicius S, Robertsson O, Kesteris U, Kalesinskas RJ, Wingstrand H. Effect of femoral head size on polyethylene wear and synovitis after total hip arthroplasty: a sonographic and radiographic study of 39 patients. Acta Orthop. 2008 Aug;79(4):489-93. doi: 10.1080/17453670710015472. PMID 18766481
- [Background] Harris WH, Muratoglu OK. A review of current cross-linked polyethylenes used in total joint arthroplasty. Clin Orthop Relat Res. 2005 Jan;(430):46-52. doi: 10.1097/01.blo.0000152603.58384.e9. PMID 15662303
- [Background] Jacobs JJ, Roebuck KA, Archibeck M, Hallab NJ, Glant TT. Osteolysis: basic science. Clin Orthop Relat Res. 2001 Dec;(393):71-7. doi: 10.1097/00003086-200112000-00008. PMID 11764373
- [Background] Doorn PF, Campbell PA, Worrall J, Benya PD, McKellop HA, Amstutz HC. Metal wear particle characterization from metal on metal total hip replacements: transmission electron microscopy study of periprosthetic tissues and isolated particles. J Biomed Mater Res. 1998 Oct;42(1):103-11. doi: 10.1002/(sici)1097-4636(199810)42:13.0.co;2-m. PMID 9740012
- [Background] Campbell DG, Field JR, Callary SA. Second-generation highly cross-linked X3 polyethylene wear: a preliminary radiostereometric analysis study. Clin Orthop Relat Res. 2010 Oct;468(10):2704-9. doi: 10.1007/s11999-010-1259-y. Epub 2010 Feb 12. PMID 20151231
- [Background] Ries MD, Pruitt L. Effect of cross-linking on the microstructure and mechanical properties of ultra-high molecular weight polyethylene. Clin Orthop Relat Res. 2005 Nov;440:149-56. doi: 10.1097/01.blo.0000185310.59202.e5. PMID 16239799
- [Background] Bitsch RG, Loidolt T, Heisel C, Ball S, Schmalzried TP. Reduction of osteolysis with use of Marathon cross-linked polyethylene. A concise follow-up, at a minimum of five years, of a previous report. J Bone Joint Surg Am. 2008 Jul;90(7):1487-91. doi: 10.2106/JBJS.F.00991. PMID 18594097
- [Background] Rohrl S, Nivbrant B, Mingguo L, Hewitt B. In vivo wear and migration of highly cross-linked polyethylene cups a radiostereometry analysis study. J Arthroplasty. 2005 Jun;20(4):409-13. doi: 10.1016/j.arth.2004.09.040. PMID 16124954
- [Background] Rohrl SM, Li MG, Nilsson KG, Nivbrant B. Very low wear of non-remelted highly cross-linked polyethylene cups: an RSA study lasting up to 6 years. Acta Orthop. 2007 Dec;78(6):739-45. doi: 10.1080/17453670710014509. PMID 18236179
- [Background] Malchau H. Revision total hip arthroplasty. Failure mechanisms and outcomes. Orthopedics. 1996 Sep;19(9):769-70. doi: 10.3928/0147-7447-19960901-17. No abstract available. PMID 8887419